CLINICAL TRIAL: NCT01149343
Title: Study of GSK2302025A Antigen-Specific Cancer Immunotherapeutic in Patients With Metastatic Melanoma
Brief Title: Evaluation of a New Vaccine Treatment for Patients With Metastatic Skin Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113173; 2009-016636-13 (EudraCT Number)
Record Dates: First submitted 2010-06-22; First posted 2010-06-23 (Estimated); Results first posted 2018-08-31 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Melanoma
Keywords: PRAME; Cancer immunotherapeutic; Malignant melanoma; ASCI (Antigen-Specific Cancer Immunotherapeutic)
MeSH Terms: conditions — Melanoma; Atypical Squamous Cells of the Cervix

ARMS (4):
- GSK2302025A Cohort 1 (Experimental): Male or female patients with histologically proven cutaneous melanoma received the investigational Low-Dose (LD) adjuvanted GSK2302025A immunotherapeutic vaccine, intramuscularly into the deltoid or lateral region of the thigh, with alternation on right or left side at each succeeding injection. Subjects received a total of 24 administrations in 4 cycles: 6 administrations given at 2 weeks intervals in cycle 1, 6 administrations given at 3 weeks intervals in cycle 2, 4 administrations given at 6 weeks intervals in cycle 3 and 4 administrations given at 3 months interval in cycle 4.
  Interventions: Biological: Immunotherapeutic GSK2302025A, different formulations
- GSK2302025A Cohort 2 (Experimental): Male or female patients with histologically proven cutaneous melanoma received the investigational Middle-Dose (MD) adjuvanted GSK2302025A immunotherapeutic vaccine, intramuscularly into the deltoid or lateral region of the thigh, with alternation on right or left side at each succeeding injection. Subjects received a total of 24 administrations in 4 cycles: 6 administrations given at 2 weeks intervals in cycle 1, 6 administrations given at 3 weeks intervals in cycle 2, 4 administrations given at 6 weeks intervals in cycle 3 and 4 administrations given at 3 months interval in cycle 4.
  Interventions: Biological: Immunotherapeutic GSK2302025A, different formulations
- GSK2302025A Cohort 3 (Experimental): Male or female patients with histologically proven cutaneous melanoma received the investigational High-Dose (HD) adjuvanted GSK2302025A immunotherapeutic vaccine, intramuscularly into the deltoid or lateral region of the thigh, with alternation on right or left side at each succeeding injection. Subjects received a total of 24 administrations in 4 cycles: 6 administrations given at 2 weeks intervals in cycle 1, 6 administrations given at 3 weeks intervals in cycle 2, 4 administrations given at 6 weeks intervals in cycle 3 and 4 administrations given at 3 months interval in cycle 4.
  Interventions: Biological: Immunotherapeutic GSK2302025A, different formulations
- GSK2302025A Cohort 4 (Experimental): In Phase 2 of the study subjects received the optimal investigational dose-level identified in Phase 1. Patients received a treatment consisting of 24 injections of the experimental GSK2302025A immunotherapeutic.
  Interventions: Biological: Immunotherapeutic GSK2302025A, different formulations

INTERVENTIONS:
Biological: Immunotherapeutic GSK2302025A, different formulations — Intramuscular administration
  Other Names: PRAME ASCI

SUMMARY:
The purpose of this clinical study is to examine the safety, immunogenicity and clinical activity of the immunotherapeutic product GSK2302025A (also referred to as recPRAME + AS15 Antigen-Specific Cancer Immunotherapeutic [ASCI]) administered as a first line treatment in patients with unresectable and progressive metastatic cutaneous melanoma.

DETAILED DESCRIPTION:
In this study, patients were to receive a maximum of 24 doses of recMAGE-A3 + AS15 according to four cycles over a period of four years. An active follow-phase (up to five years after registration into the study) was planned for all patients.

This protocol summary has been impacted by protocol amendment 3, so there will no longer be an active follow-up of patients after discontinuation or completion of the study treatment. The study will end approximately 30 days after the last dose will be administered.

In addition, no more biological samples will be collected for protocol research purposes. For each biological sample already collected in the scope of this study and not tested yet, testing will not be performed by default, except if a scientific rationale remains relevant.

Sampling for safety monitoring as per protocol will continue.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient with histologically proven cutaneous melanoma. Phase I segment: All melanoma patients with stage IV M1b and stage IV M1c including completely resected stage IV patients but with the exception of stage IV M1c disease with serum lactate dehydrogenase > 1.5 x Upper Limit of Normal or with involvement of the Central Nervous System.

   Phase II segment: All melanoma patients with measurable, unresectable stage III melanoma including in-transit metastasis (with (N3) or without (N2c) nodal metastasis) and stage IV M1a melanoma. The patient should have documented progressive disease within 12 weeks of registration into the trial. Patients with resected stage IV and with stage IV M1b or M1c disease cannot be included.
2. Written informed consent for PRAME expression screening and gene profiling on resected tumor tissue and for the complete study has been obtained from the patient prior to shipment of the sample for expression testing and prior to the performance of any other protocol-specific procedure.
3. The patient is >= 18 years old at the time of signing the first informed consent form.
4. The patient's tumor shows expression of the PRAME antigen as determined by RT-PCR analysis or any updated technique on fresh tissue sample.
5. Eastern Cooperative Oncology Group performance status of 0 or 1.
6. The patient has adequate bone marrow reserve, renal, adrenal and hepatic function as assessed by standard laboratory criteria.
7. Female patients of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as current tubal ligation, hysterectomy, ovariectomy or post-menopause.
8. Female patients of childbearing potential may be enrolled in the study, if the patient:

   * has practiced adequate contraception for 30 days prior to the study product administration, and
   * has a negative pregnancy test on the day of administration, and
   * has agreed to continue adequate contraception during the entire treatment period and for 2 months after the completion of the study product administration series.
9. In the view of the investigator, the patient can and will comply with all the requirements of the protocol.

Exclusion Criteria:

1. The patient has at any time received systemic chemotherapy, (bio)-chemotherapy or CTLA-4 monoclonal antibodies for metastatic disease.
2. The patient is scheduled to receive any other anticancer treatment, including but not limited to (bio)-chemotherapeutic or immunomodulating agents and radiotherapy.
3. The patient has received any cancer immunotherapy containing the PRAME antigen or any cancer immunotherapy for his/her metastatic disease.
4. The patient requires concomitant treatment (more than 7 consecutive days) with systemic corticosteroids or any other immunosuppressive agents.
5. Use of any investigational or non-registered product (drug or vaccine) other than the study product within the 30 days preceding the first ASCI dose injection or planned use during the study period
6. The patient has (had) previous or concomitant malignancies at other sites (including carcinoma in situ), except effectively treated non-melanoma skin cancers or carcinoma in situ of the cervix or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
7. The patient has an allergy to any component of the study investigational product or has a history of previous allergic reactions to vaccinations.
8. The patient has a history of confirmed adrenal dysfunction.
9. The patient has an autoimmune disease such as, but not limited to, multiple sclerosis, lupus, and inflammatory bowel disease.
10. The patient is known to be positive for the human immunodeficiency virus (HIV).
11. The patient has an uncontrolled bleeding disorder.
12. The patient has a family history of congenital or hereditary immunodeficiency.
13. The patient has psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures.
14. The patient has other concurrent severe medical problems, unrelated to the malignancy, that would significantly limit full compliance with the study or expose the patient to unacceptable risk.
15. For female patients: the patient is pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-07-02 (Actual); Primary Completion 2014-02-11 (Actual); Study Completion 2016-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (35):
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Prague
- France (7):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (11):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Tübingen, Baden-Wurttemberg
  - GSK Investigational Site, Nuremberg, Bavaria
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Kiel, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
- Italy (7):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Meldola (FC), Emilia-Romagna
  - GSK Investigational Site, Ravenna, Emilia-Romagna
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano (MI), Lombardy
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Słupsk
- Russia (4):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=5107

REFERENCES:
- [Derived] Gutzmer R, Rivoltini L, Levchenko E, Testori A, Utikal J, Ascierto PA, Demidov L, Grob JJ, Ridolfi R, Schadendorf D, Queirolo P, Santoro A, Loquai C, Dreno B, Hauschild A, Schultz E, Lesimple TP, Vanhoutte N, Salaun B, Gillet M, Jarnjak S, De Sousa Alves PM, Louahed J, Brichard VG, Lehmann FF. Safety and immunogenicity of the PRAME cancer immunotherapeutic in metastatic melanoma: results of a phase I dose escalation study. ESMO Open. 2016 Aug 8;1(4):e000068. doi: 10.1136/esmoopen-2016-000068. eCollection 2016. PMID 27843625

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Started (107 patients were treated, 106 patients have 1 dose of vaccine assigned in the randomization system) | 20 | 24 | 22 | 40
Completed | 0 | 0 | 0 | 0
Not Completed | 20 | 24 | 22 | 40
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 5
Not completed — Death | 10 | 13 | 18 | 18
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1
Not completed — Other | 8 | 10 | 2 | 14
Not completed — Sponsor study termination | 0 | 0 | 0 | 2
Not completed — Recurrence / Progressive disease | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4 | Total
Number analyzed (Participants) | 20 | 24 | 22 | 40 | 106
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.3 (14.9) | 60.8 (15.5) | 59.5 (15.2) | 60.7 (18.1) | 60.4 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 10 | 29 | 57
  Male | 13 | 13 | 12 | 11 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic Ancestry: White - Caucasian / European Heritage | 20 | 23 | 21 | 40 | 104
  Geographic Ancestry: Unspecified | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose-limiting Toxicity (Phase I)
Description: The dose-limiting toxicities (DLT) were defined as follows: •An Antigen-Specific Cancer Immunotherapeutic (ASCI) related or possibly ASCI related grade 3 or higher toxicity. Grade 3 myalgia, arthralgia, headache, fever, rigors/chills and fatigue (including lethargy, malaise and asthenia) persisting for 48 hours despite therapy. •An ASCI related or possibly ASCI related grade 2 or higher allergic reaction occurring within 24 hours following the ASCI administration. •An ASCI related or possibly ASCI related decrease in renal function, with a creatinine clearance lower than (<) 40 milliliters per minute (mL/min). •An ASCI-related or possibly ASCI-related symptomatic and confirmed adrenal insufficiency. The grading used was defined according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0: Grade 3 DLT = severe DLT. Related = DLT considered by investigator as possibly related to product administration.
Time Frame: During the study treatment (up to Year 4), for all patients
Population: The analysis was performed on Phase 1 subjects from the Total treated population, which included all enrolled patients who have received at least one study dose injection.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3
Number analyzed (Participants) | 20 | 24 | 22
Participants
  Patients with DLT | 0 | 1 | 1
  Patients with related DLT | 0 | 1 | 1
  Patients with severe DLT | 0 | 1 | 1
  Brain oedema | 0 | 1 | 0
  Microalbuminuria | 0 | 0 | 1
  Proteinuria | 0 | 0 | 1

2. Primary Outcome: Percentage of Patients With Anti-PReferentially Expressed Antigen of MElanoma (Anti-PRAME) Humoral Immune Response (Phase I)
Description: A seronegative/seropositive patient for anti-PRAME antibodies was a patient with antibody concentration lower (<)/ higher than or equal to (≥) cut-off level. Humoral immune response was defined as a) if baseline concentration < cut-off level: post treatment concentration ≥ cut-off level, or b) if baseline concentration ≥ cut-off level: post treatment concentration at least twice the baseline value. Cut-off values for seropositivity (by enzyme-linked immunosorbent assay [ELISA]) were 12 ELISA Units per milliliter (EL.U/mL).
Time Frame: After the administration of dose 4, at Week 8
Population: The analysis was performed on Phase 1 subjects with available results at Week 8, from the Total treated population, which included all enrolled patients who have received at least one study dose injection.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3
Number analyzed (Participants) | 13 | 13 | 17
Percentage of patients | 100 [75.3 to 100] | 100 [75.3 to 100] | 100 [80.5 to 100]

3. Primary Outcome: Number of Patients With Best Overall Response to Study Treatment (Phase II)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started). In general the patient's best response assignment depended on the achievement of both measurement and confirmation criteria. The best overall response includes the complete response (CR) defined as disappearance of all targeted/non-targeted lesions and partial response (PR) defined as at least 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD and persistence of one or more non-targeted lesion(s).
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: The analysis was performed on the Total treated population, which included all enrolled patients who have received at least one study dose injection.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  Patients with CR | 0 | 0 | 0 | 0
  Patients with PR | 0 | 0 | 0 | 4

4. Secondary Outcome: Number of Patients With Any Unsolicited Adverse Events (AEs), by Maximum Grading
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. The grading to be used by the investigators for the assessment of the severity of adverse events (AEs) was defined as the Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 (Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe or medically significant; Grade 4 = life-threatening; Grade 5 = death related to AE). Adverse Events were coded to the preferred term (PT) level by means of the Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  Grade 1 | 9 | 9 | 8 | 12
  Grade 2 | 6 | 6 | 10 | 15
  Grade 3 | 4 | 5 | 3 | 7
  Grade 4 | 1 | 1 | 0 | 3
  Grade 5 | 0 | 0 | 0 | 2

5. Secondary Outcome: Number of Patients With Serious Adverse Events (SAEs), by Maximum Grading
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity. The grading to be used by the investigators for the assessment of the severity of adverse events (AEs) was defined as the Common Terminology Criteria for Adverse Events (CTCAE), Version 4.0 (Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe or medically significant; Grade 4 = life-threatening; Grade 5 = death related to AE). SAEs were coded to the preferred term (PT) level by means of the Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  Grade 1 | 0 | 0 | 0 | 0
  Grade 2 | 0 | 0 | 1 | 0
  Grade 3 | 2 | 2 | 1 | 0
  Grade 4 | 1 | 1 | 0 | 3
  Grade 5 | 0 | 0 | 0 | 2

6. Secondary Outcome: Number of Patients With Laboratory Abnormalities Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Unknown) were compared to each baseline parameter grade (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [APTTP] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [APTTP], G0-GUnknown | 0 | 0 | 0 | 0
  [APTTP], G1-GUnknown | 0 | 0 | 0 | 0
  [APTTP], G2-GUnknown | 0 | 0 | 0 | 0
  [APTTP], G3-GUnknown | 0 | 0 | 0 | 1
  [APTTP], G4-GUnknown | 0 | 0 | 0 | 0
  [APTTP], GUknown-GUnknown | 2 | 0 | 1 | 0
  [APTTP], G0-G0 | 13 | 16 | 18 | 33
  [APTTP], G1-G0 | 2 | 3 | 1 | 3
  [APTTP], G2-G0 | 0 | 0 | 1 | 0
  [APTTP], G3-G0 | 0 | 1 | 0 | 1
  [APTTP], G4-G0 | 0 | 0 | 0 | 0
  [APTTP], GUnknown-G0 | 2 | 0 | 1 | 0
  [APTTP], G0-G1 | 0 | 1 | 0 | 1
  [APTTP], G1-G1 | 0 | 2 | 0 | 0
  [APTTP], G2-G1 | 0 | 0 | 0 | 1
  [APTTP], G3-G1 | 0 | 0 | 0 | 0
  [APTTP], G4-G1 | 0 | 0 | 0 | 0
  [APTTP], GUnknown-G1 | 0 | 1 | 0 | 0
  [APTTP], G0-G2 | 0 | 0 | 0 | 0
  [APTTP], G1-G2 | 0 | 0 | 0 | 0
  [APTTP], G2-G2 | 1 | 0 | 0 | 0
  [APTTP], G3-G2 | 0 | 0 | 0 | 0
  [APTTP], G4-G2 | 0 | 0 | 0 | 0
  [APTTP], GUknown-G2 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Patients With Laboratory Abnormal Results Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to each baseline parameter grade (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [ALT/I] and [APH/I] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 22 | 24 | 40
Participants
  [ALT/I], G0-G0 | 11 | 18 | 16 | 34
  [ALT/I], G1-G0 | 4 | 4 | 5 | 1
  [ALT/I], G2-G0 | 0 | 0 | 0 | 1
  [ALT/I], G3-G0 | 0 | 0 | 0 | 0
  [ALT/I], G4-G0 | 0 | 0 | 0 | 0
  [ALT/I], GUknown-G0 | 2 | 0 | 1 | 0
  [ALT/I], G0-G1 | 0 | 2 | 0 | 1
  [ALT/I], G1-G1 | 3 | 0 | 0 | 3
  [ALT/I], G2-G1 | 0 | 0 | 0 | 0
  [ALT/I], G3-G1 | 0 | 0 | 0 | 0
  [ALT/I], G4-G1 | 0 | 0 | 0 | 0
  [ALT/I], GUknown-G1 | 0 | 0 | 0 | 0
  [APH/I], G0-G0 | 16 | 20 | 15 | 33
  [APH/I], G1-G0 | 1 | 3 | 5 | 5
  [APH/I], G2-G0 | 0 | 0 | 1 | 1
  [APH/I], G3-G0 | 0 | 0 | 0 | 0
  [APH/I], G4-G0 | 0 | 0 | 0 | 0
  [APH/I], GUknown-G0 | 2 | 0 | 1 | 0
  [APH/I], G0-G1 | 0 | 0 | 0 | 0
  [APH/I], G1-G1 | 0 | 0 | 0 | 1
  [APH/I], G2-G1 | 0 | 1 | 0 | 0
  [APH/I], G3-G1 | 0 | 0 | 0 | 0
  [APH/I], G4-G1 | 0 | 0 | 0 | 0
  [APH/I], GUknokwn-G1 | 0 | 0 | 0 | 0
  [APH/I], G0-G2 | 0 | 0 | 0 | 0
  [APH/I], G1-G2 | 0 | 0 | 0 | 0
  [APH/I], G2-G2 | 0 | 0 | 0 | 0
  [APH/I], G3-G2 | 1 | 0 | 0 | 0
  [APH/I], G4-G2 | 0 | 0 | 0 | 0
  [APH/I], GUknown-G2 | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Patients With Hematological and Biochemical Abnormalities Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to baseline parameter grades (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [AN], [AST/I] and [CRE/I] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [AN], G0-G0 | 12 | 10 | 10 | 21
  [AN], G1-G0 | 1 | 6 | 5 | 12
  [AN], G2-G0 | 0 | 0 | 1 | 3
  [AN], G3-G0 | 1 | 0 | 0 | 0
  [AN], G4-G0 | 0 | 0 | 0 | 0
  [AN], GUknown-G0 | 1 | 0 | 1 | 0
  [AN], G0-G1 | 2 | 1 | 0 | 0
  [AN], G1-G1 | 2 | 5 | 5 | 4
  [AN], G2-G1 | 0 | 1 | 0 | 0
  [AN], G3-G1 | 0 | 1 | 0 | 0
  [AN], G4-G1 | 0 | 0 | 0 | 0
  [AN], GUnknown-G1 | 1 | 0 | 0 | 0
  [AST/I], G0-G0 | 13 | 18 | 17 | 36
  [AST/I], G1-G0 | 3 | 6 | 4 | 2
  [AST/I], G2-G0 | 0 | 0 | 0 | 0
  [AST/I], G3-G0 | 0 | 0 | 0 | 0
  [AST/I], G4-G0 | 0 | 0 | 0 | 0
  [AST/I], GUnknown-G0 | 1 | 0 | 1 | 0
  [AST/I], G0-G1 | 1 | 0 | 0 | 0
  [AST/I], G1-G1 | 1 | 0 | 0 | 2
  [AST/I], G2-G1 | 0 | 0 | 0 | 0
  [AST/I], G3-G1 | 0 | 0 | 0 | 0
  [AST/I], G4-G1 | 0 | 0 | 0 | 0
  [AST/I], GUnknown-G1 | 1 | 0 | 0 | 0
  [BB/I], G0-G0 | 16 | 21 | 19 | 38
  [BB/I], G1-G0 | 1 | 2 | 1 | 0
  [BB/I], G2-G0 | 1 | 0 | 0 | 0
  [BB/I], G3-G0 | 0 | 0 | 0 | 0
  [BB/I], G4-G0 | 0 | 0 | 0 | 0
  [BB/I], GUnknown-G0 | 2 | 0 | 1 | 0
  [BB/I], G0-G1 | 0 | 0 | 0 | 0
  [BB/I], G1-G1 | 0 | 1 | 1 | 1
  [BB/I], G2-G1 | 0 | 0 | 0 | 1
  [BB/I], G3-G1 | 0 | 0 | 0 | 0
  [BB/I], G4-G1 | 0 | 0 | 0 | 0
  [BB/I], GUnknown-G1 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Patients With Laboratory Hematological and Biochemical Abnormalities Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to baseline parameter grades (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [CRE/I] and [GGT/I] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [CRE/I], G0-G0 | 20 | 22 | 20 | 33
  [CRE/I], G1-G0 | 0 | 0 | 1 | 6
  [CRE/I], G2-G0 | 0 | 0 | 0 | 0
  [CRE/I], G3-G0 | 0 | 0 | 0 | 0
  [CRE/I], G4-G0 | 0 | 0 | 0 | 0
  [CRE/I], GUnknown-G0 | 0 | 0 | 0 | 0
  [CRE/I], G0-G1 | 0 | 0 | 0 | 0
  [CRE/I], G1-G1 | 0 | 1 | 1 | 0
  [CRE/I], G2-G1 | 0 | 0 | 0 | 0
  [CRE/I], G3-G1 | 0 | 0 | 0 | 0
  [CRE/I], G4-G1 | 0 | 0 | 0 | 0
  [CRE/I], GUnknown-G1 | 0 | 0 | 0 | 0
  [CRE/I], G0-G2 | 0 | 0 | 0 | 0
  [CRE/I], G1-G2 | 0 | 0 | 0 | 0
  [CRE/I], G2-G2 | 0 | 1 | 0 | 1
  [CRE/I], G3-G2 | 0 | 0 | 0 | 0
  [CRE/I], G4-G2 | 0 | 0 | 0 | 0
  [CRE/I], GUknown-G2 | 0 | 0 | 0 | 0
  [GGT/I], G0-G0 | 10 | 17 | 14 | 30
  [GGT/I], G1-G0 | 1 | 1 | 1 | 4
  [GGT/I], G2-G0 | 2 | 2 | 1 | 0
  [GGT/I], G3-G0 | 0 | 0 | 0 | 0
  [GGT/I], G4-G0 | 0 | 0 | 0 | 1
  [GGT/I], GUnknown-G0 | 1 | 0 | 1 | 0
  [GGT/I], G0-G1 | 2 | 1 | 1 | 1
  [GGT/I], G1-G1 | 0 | 1 | 1 | 3
  [GGT/I], G2-G1 | 1 | 1 | 0 | 0
  [GGT/I], G3-G1 | 0 | 0 | 1 | 0
  [GGT/I], G4-G1 | 0 | 0 | 0 | 0
  [GGT/I], GUnknown-G1 | 1 | 0 | 0 | 0
  [GGT/I], G0-G2 | 0 | 0 | 0 | 0
  [GGT/I], G1-G2 | 0 | 1 | 0 | 0
  [GGT/I], G2-G2 | 0 | 0 | 0 | 0
  [GGT/I], G3-G2 | 1 | 0 | 2 | 0
  [GGT/I], G4-G2 | 0 | 0 | 0 | 0
  [GGT/I], GUnknown-G2 | 1 | 0 | 0 | 0
  [GGT/I], G0-G3 | 0 | 0 | 0 | 0
  [GGT/I], G1-G3 | 0 | 0 | 0 | 0
  [GGT/I], G2-G3 | 0 | 0 | 0 | 0
  [GGT/I], G3-G3 | 0 | 0 | 0 | 1
  [GGT/I], G4-G3 | 0 | 0 | 0 | 0
  [GGT/I], GUnknown-G3 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Patients With Lab Hematological and Biochemical Abnormalities Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to each baseline parameter grade (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [Hgb/I] and [HYP] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [Hgb/I], G0-G0 | 16 | 24 | 21 | 37
  [Hgb/I], G1-G0 | 0 | 0 | 0 | 2
  [Hgb/I], G2-G0 | 0 | 0 | 0 | 0
  [Hgb/I], G3-G0 | 0 | 0 | 0 | 0
  [Hgb/I], G4-G0 | 0 | 0 | 0 | 0
  [Hgb/I], GUnknown-G0 | 2 | 0 | 1 | 0
  [Hgb/I], G0-G1 | 0 | 0 | 0 | 0
  [Hgb/I], G1-G1 | 1 | 0 | 0 | 0
  [Hgb/I], G2-G1 | 0 | 0 | 0 | 1
  [Hgb/I], G3-G1 | 0 | 0 | 0 | 0
  [Hgb/I], G4-G1 | 0 | 0 | 0 | 0
  [Hgb/I], GUnknown-G1 | 0 | 0 | 0 | 0
  [Hgb/I], G0-G2 | 0 | 0 | 0 | 0
  [Hgb/I], G1-G2 | 1 | 0 | 0 | 0
  [Hgb/I], G2-G2 | 0 | 0 | 0 | 0
  [Hgb/I], G3-G2 | 0 | 0 | 0 | 0
  [Hgb/I], G4-G2 | 0 | 0 | 0 | 0
  [Hgb/I], GUnknown-G2 | 0 | 0 | 0 | 0
  [HYP], G0-G0 | 13 | 17 | 18 | 30
  [HYP], G1-G0 | 2 | 5 | 2 | 5
  [HYP], G2-G0 | 0 | 1 | 0 | 1
  [HYP], G3-G0 | 0 | 0 | 0 | 0
  [HYP], G4-G0 | 0 | 0 | 0 | 0
  [HYP], GUnknown-G0 | 3 | 0 | 2 | 0
  [HYP], G0-G1 | 0 | 0 | 0 | 0
  [HYP], G1-G1 | 1 | 1 | 0 | 3
  [HYP], G2-G1 | 1 | 0 | 0 | 0
  [HYP], G3-G1 | 0 | 0 | 0 | 0
  [HYP], G4-G1 | 0 | 0 | 0 | 0
  [HYP], GUnknown-G1 | 0 | 0 | 0 | 0
  [HYP], G0-G3 | 0 | 0 | 0 | 1
  [HYP], G1-G3 | 0 | 0 | 0 | 0
  [HYP], G2-G3 | 0 | 0 | 0 | 0
  [HYP], G3-G3 | 0 | 0 | 0 | 0
  [HYP], G4-G3 | 0 | 0 | 0 | 0
  [HYP], GUnknown-G3 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Patients With Abnormal Hematological and Biochemical Results Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [ NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to each baseline parameter grade (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [LYMC/D] and [LYMC/I] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [LYMC/D], G0-G0 | 10 | 14 | 14 | 28
  [LYMC/D], G1-G0 | 3 | 4 | 3 | 4
  [LYMC/D], G2-G0 | 1 | 1 | 0 | 0
  [LYMC/D], G3-G0 | 0 | 0 | 0 | 0
  [LYMC/D], G4-G0 | 0 | 0 | 0 | 0
  [LYMC/D], GUnknown-G0 | 0 | 0 | 1 | 0
  [LYMC/D], G0-G1 | 0 | 1 | 1 | 2
  [LYMC/D], G1-G1 | 3 | 3 | 2 | 5
  [LYMC/D], G2-G1 | 1 | 0 | 0 | 0
  [LYMC/D], G3-G1 | 0 | 0 | 0 | 0
  [LYMC/D], G4-G1 | 0 | 0 | 0 | 0
  [LYMC/D], GUnknown-G1 | 1 | 1 | 0 | 0
  [LYMC/D], G0-G2 | 0 | 0 | 0 | 0
  [LYMC/D], G1-G2 | 0 | 0 | 1 | 0
  [LYMC/D], G2-G2 | 0 | 0 | 0 | 1
  [LYMC/D], G3-G2 | 0 | 0 | 0 | 0
  [LYMC/D], G4-G2 | 0 | 0 | 0 | 0
  [LYMC/D], GUnknown-G2 | 0 | 0 | 0 | 0
  [LYMC/D], G0-G3 | 0 | 0 | 0 | 0
  [LYMC/D], G1-G3 | 0 | 0 | 0 | 0
  [LYMC/D], G2-G3 | 0 | 0 | 0 | 0
  [LYMC/D], G3-G3 | 0 | 0 | 0 | 0
  [LYMC/D], G4-G3 | 0 | 0 | 0 | 0
  [LYMC/D], GUnknown-G3 | 1 | 0 | 0 | 0
  [LYMC/I], G0-G0 | 16 | 23 | 21 | 40
  [LYMC/I], G1-G0 | 0 | 0 | 0 | 0
  [LYMC/I], G2-G0 | 2 | 0 | 0 | 0
  [LYMC/I], G3-G0 | 0 | 0 | 0 | 0
  [LYMC/I], G4-G0 | 0 | 0 | 0 | 0
  [LYMC/I], GUnknown-G0 | 2 | 1 | 1 | 0

12. Secondary Outcome: Number of Patients With Abnormal Hematological and Biochemical Laboratory Results Versus Baseline, by Maximum Grading
Description: Laboratory abnormalities belong to hematological and biochemical parameters such as: activated partial thromboplastin time prolonged [APTTP], alanine aminotransferase increased [ALT/I], alkaline phoshatase increased [APH/I], anemia [AN], asparatate aminostransferase increased [AST/I], blood bilirubin increased [BB/I], creatinine increased [CRE/I], gamma glumatymtransferase increased [GGT/I], hemoglobin increased [Hgb/I], hypoalbuminemia [HYP], lymphocyte count decreased [LYMC/D], lymphocyte count increased [LYMC/I], neutrophil count decreased [NEUC/D], platelet count decreased [PLA/D], white blood cell decreased [WBC/D]. Parameter grades (G0,1,2,3,4,Uknown) were compared to each baseline parameter grades (GUnknown,0,1,2,3), as defined by the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of May 28, 2009 [http://evs.nci.nih.gov/ftp1/CTCAE]. This endpoint presents values for [NEUC/D], [PLA/D] and [WBC/D] grading versus baseline parameter grading.
Time Frame: During the entire study period - up to Year 4 + 1 month post last study treatment administration
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  [NEUC/D], G0-G0 | 17 | 21 | 21 | 39
  [NEUC/D], G1-G0 | 1 | 2 | 0 | 0
  [NEUC/D], G2-G0 | 0 | 0 | 0 | 0
  [NEUC/D], G3-G0 | 0 | 0 | 0 | 0
  [NEUC/D], G4-G0 | 0 | 0 | 0 | 0
  [NEUC/D], GUnknown-G0 | 2 | 1 | 1 | 0
  [NEUC/D], G0-G1 | 0 | 0 | 0 | 0
  [NEUC/D], G1-G1 | 0 | 0 | 0 | 1
  [NEUC/D], G2-G1 | 0 | 0 | 0 | 0
  [NEUC/D], G3-G1 | 0 | 0 | 0 | 0
  [NEUC/D], G4-G1 | 0 | 0 | 0 | 0
  [NEUC/D], GUnknown-G1 | 0 | 0 | 0 | 0
  [PLA/D], G0-G0 | 17 | 24 | 20 | 38
  [PLA/D], G1-G0 | 1 | 0 | 0 | 2
  [PLA/D], G2-G0 | 0 | 0 | 0 | 0
  [PLA/D], G3-G0 | 0 | 0 | 0 | 0
  [PLA/D], G4-G0 | 0 | 0 | 0 | 0
  [PLA/D], GUnknown-G0 | 2 | 0 | 1 | 0
  [PLA/D], G0-G1 | 0 | 0 | 0 | 0
  [PLA/D], G1-G1 | 0 | 0 | 1 | 0
  [PLA/D], G2-G1 | 0 | 0 | 0 | 0
  [PLA/D], G3-G1 | 0 | 0 | 0 | 0
  [PLA/D], G4-G1 | 0 | 0 | 0 | 0
  [PLA/D], GUnknown-G1 | 0 | 0 | 0 | 0
  [WBC/D], G0-G0 | 14 | 21 | 19 | 34
  [WBC/D], G1-G0 | 2 | 1 | 1 | 3
  [WBC/D], G2-G0 | 0 | 0 | 0 | 0
  [WBC/D], G3-G0 | 0 | 0 | 0 | 0
  [WBC/D], G4-G0 | 0 | 0 | 0 | 0
  [WBC/D], GUnknown-G0 | 2 | 0 | 1 | 0
  [WBC/D], G0-G1 | 1 | 0 | 0 | 2
  [WBC/D], G1-G1 | 1 | 2 | 1 | 1
  [WBC/D], G2-G1 | 0 | 0 | 0 | 0
  [WBC/D], G3-G1 | 0 | 0 | 0 | 0
  [WBC/D], G4-G1 | 0 | 0 | 0 | 0
  [WBC/D], GUnknown-G1 | 0 | 0 | 0 | 0

13. Secondary Outcome: Percentage of Patients With Anti-PRAME Cellular (T-cell) Response (Phase I)
Description: Cellular response was defined as: Geometric Mean Response (GMR) above the 2.68 cut-off value and at least a four-fold increase of PRAME- specific Cluster of Differentiation (CD) 4/8 T-cells. Considering that 2 studies failed to demonstrate clinical efficacy of recombinant protein based cancer vaccines, GSK decided in 2014 to stop the development and to stop recruitment in all the ongoing clinical studies. The decision was made to end the study (i.e., stopping patient enrollment, follow-ups, sample collection and analysis of samples for research purposes). Patients still on treatment at the time of the protocol amendment were offered to continue the administration of the study treatment until the last dose or until recurrence, whichever came first, or until the patient or the investigator decided to stop the study treatment. No further active protocol visit/contact was performed except for the concluding visit at Week 199, 30 days after the last treatment administration.
Time Frame: Up to Data Lock Point at Week 8
Population: The analysis was performed on the Phase 1 subjects with available results up to Week 8, from the Total treated population, which included all enrolled patients who have received at least one study dose injection.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3
Number analyzed (Participants) | 8 | 11 | 14
Percentage of patients
  Patients with CD4 pre+post-administration results | 100 [63.1 to 100] | 100 [71.5 to 100] | 100 [76.8 to 100]
  Responders CD4 | 75.0 [34.9 to 96.8] | 45.5 [16.7 to 76.6] | 57.1 [28.9 to 82.3]
  Patients with CD8 pre+post-administration results: number analyzed (Participants) | 8 | 9 | 8
  Patients with CD8 pre+post-administration results | 100 [63.1 to 100] | 100 [66.4 to 100] | 100 [63.1 to 100]
  Responders CD8: number analyzed (Participants) | 8 | 9 | 8
  Responders CD8 | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 33.6] | 0.0 [0.0 to 36.9]

14. Secondary Outcome: Number of Patients With Anti-PRAME Humoral Immune Response (Phase I & II)
Description: A seropositive patient was a patient whose anti-PRAME antibody concentration was greater than or equal to (≥) the assay cut-off value of 12 ELISA units per milliliter (EL.U/mL). A seronegative patient was defined as a patient whose pre-treatment antibody concentration was below (<) the cut-off value. An anti-PRAME antibody responder was defined as: For a seronegative patient: a post-treatment antibody concentration ≥ the cut-off value; For a seropositive patient: a post-treatment antibody concentration ≥ twice the pre-treatment antibody concentration.
Time Frame: At Weeks 0, 4, 8, 10, 12, 29, 51, 75, 99, 123, 147 and conclusion visit at 30 days post last treatment administration (Week 199) for each patient
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  anti-PRAME,Week 0 | 0 | 0 | 0 | 2
  anti-PRAME, Week 4: number analyzed (Participants) | 15 | 18 | 21 | 36
  anti-PRAME, Week 4 | 11 | 14 | 18 | 33
  anti-PRAME, Week 8: number analyzed (Participants) | 14 | 13 | 21 | 33
  anti-PRAME, Week 8 | 14 | 13 | 21 | 33
  anti-PRAME, Week 10: number analyzed (Participants) | 10 | 12 | 19 | 33
  anti-PRAME, Week 10 | 10 | 12 | 19 | 33
  anti-PRAME, Week 12: number analyzed (Participants) | 9 | 9 | 16 | 28
  anti-PRAME, Week 12 | 9 | 9 | 16 | 28
  anti-PRAME, Week 29: number analyzed (Participants) | 2 | 4 | 5 | 13
  anti-PRAME, Week 29 | 2 | 4 | 5 | 13
  anti-PRAME, Week 51: number analyzed (Participants) | 1 | 3 | 3 | 7
  anti-PRAME, Week 51 | 1 | 3 | 3 | 7
  anti-PRAME, Week 75: number analyzed (Participants) | 2 | 2 | 2 | 1
  anti-PRAME, Week 75 | 2 | 2 | 2 | 1
  anti-PRAME, Week 99: number analyzed (Participants) | 2 | 2 | 2 | 0
  anti-PRAME, Week 99 | 2 | 2 | 2 | 0
  anti-PRAME, Week 123: number analyzed (Participants) | 1 | 1 | 1 | 0
  anti-PRAME, Week 123 | 1 | 1 | 1 | 0
  anti-PRAME, Week 147: number analyzed (Participants) | 1 | 0 | 0 | 0
  anti-PRAME, Week 147 | 1 | 0 | 0 | 0
  anti-PRAME, Week 199: number analyzed (Participants) | 6 | 12 | 8 | 23
  anti-PRAME, Week 199 | 6 | 12 | 8 | 23

15. Secondary Outcome: Number of Patients With Stable Disease (SD), Progressive Disease (PD), Mixed Response (MR) (Phase I & II)
Description: Tumor response was assessed by the Response Evaluation Criteria In Solid Tumors (RECIST), where stable disease for target lesions refers to neither enough shrinkage to qualify for complete response nor sufficient increase to qualify for progressive disease taking as references the smallest sum longest diameter (LD) since the treatment started. For non-targeted lesions it refers to persistence of one or more non-target lesions. Progressive disease is related to a clear increase of diameters of lesions taking as references the smallest diameters recorded since the treatment started OR the appearance of one or more new lesions OR both of these.
Time Frame: At 30 days after the last treatment administration for each patient (Week 199)
Population: The analysis was performed on the Total Vaccinated Cohort, which included all enrolled patients who have received at least one study dose injection.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  Complete response | 0 | 0 | 0 | 0
  Partial response | 0 | 0 | 0 | 4
  Stable disease | 2 | 1 | 1 | 1
  Stable Disease/Progressive disease | 0 | 1 | 1 | 3
  Progressive disease | 9 | 18 | 15 | 31
  Non Evaluable | 2 | 1 | 0 | 1
  Missing Best overall response | 7 | 3 | 5 | 0
  Disease control: Yes | 2 | 2 | 2 | 8
  Disease control: No | 18 | 22 | 20 | 32

16. Secondary Outcome: Number of Patients With Best Overall Response, Including Mixed Response (MxR) and Slow Progressive Disease (SPD) Criteria (Phase I & II)
Description: Tumor response was assessed by the RECIST criteria, where SD for target lesions refers to neither enough shrinkage to qualify for CR nor sufficient increase to qualify for PD taking as references the smallest sum longest diameter (LD) since the treatment started. For non-targeted lesions it refers to persistence of one or more nom-target lesions. Progressive disease is related to a clear increase of diameters of lesions taking as references the smallest diameters recorded since the treatment started OR the appearance of one or more new lesions OR both of these. Mixed response is defined as at least 30% decrease in the LD occurring in at least one target lesion recorded and measured at baseline. Such response occurring in otherwise SD or PD status of the LD of target lesions were classified as "SD with target lesion regression" or "PD with target lesion regression", respectively. New lesion(s) in otherwise PR status of the LD of target lesions were "PR with new lesion".
Time Frame: At 30 days after the last treatment administration for each patient (Week 199)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Participants
  PR | 0 | 0 | 0 | 0
  CR | 0 | 0 | 0 | 4
  MxR: SD with target lesion regression | 0 | 0 | 0 | 0
  MxR: PD with target lesion regression | 2 | 2 | 2 | 3
  MxR: PR with new lesion | 0 | 0 | 1 | 0
  SD/PR | 0 | 1 | 1 | 3
  SD without mixed response | 2 | 0 | 1 | 1
  PD with SPD criteria | 3 | 5 | 4 | 19
  PD without SPD/MxR | 4 | 12 | 8 | 9
  Non Evaluable | 2 | 1 | 0 | 1
  Missing Best overall response | 7 | 3 | 5 | 0

17. Secondary Outcome: Anti-Protein D Humoral Response (Phase I & II)
Description: Analysis of immunogenicity for anti-PD antibodies was not performed, following negative results to the NCT00480025 study which assessed another study product from same technology platform. For this study, the main analysis of the dose-escalation Phase I segment was performed according to protocol when all patients enrolled in the Phase I segment had received the first 4 treatment doses and had completed Week 8. The main analysis of the Phase II segment was performed according to protocol when all patients had either completed the treatment until the end of Cycle 3 or had been withdrawn from the study treatment, with the exception of anti-PD antibody responses and PRAME-specific cellular responses which were not yet performed. All samples that had been collected but not yet tested were not tested by default, except if a scientific rationale remained relevant.
Time Frame: At Week 0, 4, 8, 12, 29, 51, 75, 99, 123, 147, 30 days after the last treatment administration for each patient (Week 199), with follow-up, 3, 6, 9 and 12 months after concluding visit
Population: This analysis was not performed.
Groups:
- GSK2302025A Cohort 1: Subjects will receive investigational dose-level A (different from dose-levels B and C). Patients will receive a treatment consisting of 24 injections of the experimental GSK2302025A immunotherapeutic
- GSK2302025A Cohort 2: Subjects will receive investigational dose-level B (different from dose-levels A and C). Patients will receive a treatment consisting of 24 injections of the experimental GSK2302025A immunotherapeutic
- GSK2302025A Cohort 3: Subjects will receive investigational dose-level C (different from dose-levels A and B). Patients will receive a treatment consisting of 24 injections of the experimental GSK2302025A immunotherapeutic
- GSK2302025A Cohort 4: In Phase 2 of the study subjects will receive the optimal investigational dose-level identified in Phase 1. Patients will receive a treatment consisting of 24 injections of the experimental GSK2302025A immunotherapeutic
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Anti-Cytosine Phosphate Guanosine Oligodeoxynucleotide (CpG) Humoral Response (Phase I & II)
Description: Analysis of immunogenicity for anti-CpG antibodies was not performed, following negative results to the NCT00480025 study which assessed another study product from same technology platform. For this study, the main analysis of the dose-escalation Phase I segment was performed according to protocol when all patients enrolled in the Phase I segment had received the first 4 treatment doses and had completed Week 8. The main analysis of the Phase II segment was performed according to protocol when all patients had either completed the treatment until the end of Cycle 3 or had been withdrawn from the study treatment, with the exception of anti-CpG antibody responses and PRAME-specific cellular responses which were not yet performed. All samples that had been collected but not yet tested were not tested by default, except if a scientific rationale remained relevant.
Time Frame: as for outcome 17
Population: This analysis was not performed.
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

19. Secondary Outcome: Time to Treatment Failure, Progression Free Survival and Overall Survival (Phase I & II)
Description: Time to treatment failure (TTF) was defined as the time from first administration of study product until the date of the last administration of the product, irrespective of the reason for study treatment discontinuation. Progression-free survival (PFS) was defined as the time from first adminsitration of study product until the date of either disease progression or death (for whatever reason), whichever comes first. Overall survival (OS) was defined as the time from first administration of study product until death.
Time Frame: Up to concluding visit, at Week 199
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 20 | 24 | 22 | 40
Months
  TTF | 2.3 [1.0 to 4.9] | 2.3 [1.3 to 4.2] | 3.0 [2.3 to 4.9] | 4.6 [2.7 to 5.3]
  PFS | 2.7 [1.4 to 2.9] | 2.7 [1.0 to 2.8] | 2.8 [2.1 to 2.9] | 2.8 [2.7 to 3.3]
  OS | 17.0 [8.1 to NA] — The upper limit of the 95% confidence interval for this group was below the limit of detection. | 11.5 [7.3 to NA] — The upper limit of the 95% confidence interval for this group was below the limit of detection. | 10.8 [8.4 to 25.5] | 23.0 [15.5 to NA] — The upper limit of the 95% confidence interval for this group was below the limit of detection.

20. Secondary Outcome: Duration of Response for Patients With CR, PR and SD or SD/PR Status (Phase II)
Description: This analysis was not performed following negative results to the NCT00480025 study which assessed another study product from same technology platform. For this study, the main analysis of the dose-escalation Phase I segment was performed according to protocol when all patients enrolled in the Phase I segment had received the first 4 treatment doses and had completed Week 8. The main analysis of the Phase II segment was performed according to protocol when all patients had either completed the treatment until the end of Cycle 3 or had been withdrawn from the study treatment, with the exception of anti-CpG/anti-PD antibody responses and PRAME-specific cellular responses which were not yet performed. All samples that had been collected but not yet tested were not tested by default, except if a scientific rationale remained relevant.
Time Frame: Up to concluding visit, at Week 199
Population: This analysis was not performed.
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Unsolicited AEs and serious adverse events (SAEs): from study start (Day 0) up to the concluding visit, at Month 49 (Week 199).
Arm/Group | GSK2302025A Cohort 1 | GSK2302025A Cohort 2 | GSK2302025A Cohort 3 | GSK2302025A Cohort 4
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/24 | 0/22 | 2/40
Serious Adverse Events (participants affected / at risk) | 3/20 | 3/24 | 2/22 | 5/40
Other Adverse Events (participants affected / at risk) | 19/20 | 21/24 | 21/22 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2302025A Cohort 1 (N=20) | GSK2302025A Cohort 2 (N=24) | GSK2302025A Cohort 3 (N=22) | GSK2302025A Cohort 4 (N=40)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK2302025A Cohort 1 (N=20) | GSK2302025A Cohort 2 (N=24) | GSK2302025A Cohort 3 (N=22) | GSK2302025A Cohort 4 (N=40)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Administration site pain (General disorders) | 0 (0) | 1 (2) | 1 (2) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Arteriosclerosis moenckeberg-type (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (24) | 1 (1) | 6 (7)
Asthenia (General disorders) | 2 (2) | 0 (0) | 6 (21) | 13 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 2 (2)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 1 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Catheter placement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (6) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 4 (10) | 1 (2) | 4 (14) | 8 (14)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 3 (3)
Cortisol decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cortisol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (6) | 0 (0) | 4 (4)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 2 (8) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 1 (1) | 1 (1) | 5 (7)
Dissociation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (2) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Fatigue (General disorders) | 5 (10) | 7 (36) | 6 (10) | 7 (12)
Feeling cold (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Glucocorticoid deficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 6 (12) | 5 (43) | 4 (9) | 7 (12)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hyperplasia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (3) | 2 (2)
Hyperthermia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 4 (18) | 6 (11) | 7 (16) | 13 (29)
Injection site erythema (General disorders) | 3 (13) | 7 (17) | 7 (14) | 8 (18)
Injection site oedema (General disorders) | 0 (0) | 1 (3) | 2 (4) | 1 (1)
Injection site pain (General disorders) | 9 (39) | 10 (32) | 12 (51) | 24 (90)
Injection site pruritus (General disorders) | 2 (2) | 2 (2) | 1 (8) | 0 (0)
Injection site reaction (General disorders) | 5 (6) | 4 (8) | 2 (5) | 2 (3)
Injection site swelling (General disorders) | 0 (0) | 1 (4) | 2 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (3)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (5) | 1 (1) | 5 (5)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (8) | 2 (2) | 11 (14)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0) | 3 (4) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (13) | 2 (3) | 8 (9)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (2) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (2)
Pyrexia (General disorders) | 6 (20) | 8 (22) | 5 (8) | 22 (86)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 4 (8) | 0 (0) | 5 (5)
Atrial fibrillation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Antinuclear antibody increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactic acid increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercreatinaemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Administration site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mood altered (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Albuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphostasis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
As a consequence of the decision to stop the study, not all data are available for a full final analysis as originally planned. Analyses are merely descriptive and the results are presented as an abridged study report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.